CLINICAL TRIAL: NCT02975752
Title: Rapid and Highly Sensitive EGFRdelEx19 and KRAS Exon 2 Mutation Detection in EBUS-TBNA Specimen of Lymph Node Metastases From Patients With Lung Adenocarcinoma
Brief Title: EGFRdelEx19 and KRAS Exon 2 Mutation Detection in EBUS-TBNA
Acronym: EGFRdelEx19
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Filiz Oezkan, Dr. med. Filiz Özkan, University Hospital, Essen
Other Study IDs: EGFRdelEx 19 KRAS Exon 2
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Lung Adenocarcinoma Metastatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — EBUS-TBNA specimen of lymph nodes and primary tumor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: LC-RT-PCR and NGS — highly sensitive PCR vs. multiplex targeted-resequencing

SUMMARY:
First-line treatment with afatinib prolongs overall survival in patients with metastatic non-small-cell lung cancer (NSCLC) harboring EGFR exon 19 deletion mutations. Conversely, somatic KRAS mutations are negative predictors for benefit from EGFR-targeting agents. In this study we want to compare a new highly sensitive method for the detection of EGFRdelEx19 and KRAS Exon 2 with targeted-resequencing multiplex-PCR (NGS).

DETAILED DESCRIPTION:
First-line treatment with afatinib prolongs overall survival in patients with metastatic non-small-cell lung cancer (NSCLC) harboring EGFR exon 19 deletion mutations. Conversely, somatic KRAS mutations are negative predictors for benefit from EGFR-targeting agents. Rapid availability of these biomarker results is mandatory to prevent delayed or inferior treatments.

Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) is well-established for lung cancer diagnosis and staging. Next generation sequencing (NGS) via targeted resequencing allows simultaneous interrogation for multiple mutations, but has its limitations based on the amount of tumor tissue required and assay times. RT-PCR using Light-Cycler technology (LC-RTPCR) is a rapid and sensitive assay to detect somatic mutations in various tissues from NSCLC patients. The study's aim was to analyze if LC-RTPCR is feasible for rapid EGFRdelEx19 and KRAS Exon 2 mutation detection in EBUS-TBNA samples and to compare results with results obtained via standard NGS mutation analyses.

ELIGIBILITY:
Inclusion Criteria:

* lung adenocarcinoma positive EBUS-TBNA specimen

Exclusion Criteria:

* other diagnosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with suspected lung cancer on the chest CT-scan images receiving EBUS-TBNA (endobronchial ultrasound-guided transbronchial needle aspiration) for clinical pre-treatment workup of mediastinal and hilar lymph nodes
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
detection of mutations | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Özkan, MD, Principal Investigator — Department of Interventional Pneumology

IPD SHARING:
Plan to Share IPD: No